CLINICAL TRIAL: NCT01667510
Title: Effect of Cardio Mato (Grade A Lyc-O-Mato, a Tomato Extracted Lycopene) on Blood Pressure and Serum Lycopene, Phytofluene, and Phytoene Levels in Pre-hypertensive Otherwise Healthy Subjects
Brief Title: Effect of Cardio Mato (Grade A Lyc-O-Mato, a Tomato Extracted Lycopene) on Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LycoRed Ltd. (Industry)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Lyc-2012-01
Record Dates: First submitted 2012-08-12; First posted 2012-08-17 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2012-08

CONDITIONS: Prehypertension
Keywords: Prehypertension; anti oxidation; lycopene
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardio Mato (Experimental): Soft gel capsule for oral use (Grade A Lyc-O-Mato, a tomato extracted lycopene)
  Interventions: Dietary Supplement: Cardio Mato
- Placebo (Placebo Comparator): Soft gel capsule without test material, for oral use
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cardio Mato — Soft gel capsule for oral use
  Arms: Cardio Mato
Dietary Supplement: Placebo — Soft gel capsule without test material
  Arms: Placebo

SUMMARY:
The hypothesis of the study is that supplementation with Cardio Mato (a Tomato Extracted Lycopene)for 12 weeks will decrease the blood pressure of subjects with prehypertension compared to Placebo.

DETAILED DESCRIPTION:
Blood-pressure reading of 140/90 mmHg (systolic/diastolic pressure) are typically regarded as having high blood pressure as defined in the most recent guidelines. From a physiological perspective, the regulation of blood pressure is a complicated process involving different biological systems and a number of feedback systems, including the nervous system, hormones, control of body fluid and regulators within the vessels themselves. In 90-95% of patients with high blood pressure the cause is unknown, whereas the remaining 5-10% may have secondary hypertension related to congenital heart defects, certain cancers or kidney abnormalities. Prehypertension [systolic blood pressure (SBP) 120-139 mm Hg, diastolic blood pressure (DBP) 80-89 mm Hg] is considered a precursor of hypertension and has been associated with an increased risk of up to 3.5 times in cardiovascular morbidity and mortality later in life.

According the report of the Joint National Committee on High Blood Pressure (JNC 7) and other international guidelines, weight control, reduced intake of salt and reduced alcohol consumption, as well as increase of potassium are recommend nutritional approaches to prevent and treat hypertension. In observational studies significant inverse association between high blood pressure and vegetarian diet rich in fibers, magnesium, potassium, calcium and protein have been reported. In addition various studies demonstrated the ability of antioxidant vitamins of natural origin to improve vascular function.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18-65, both inclusive
2. Established Pre-hypertension defined as: Mean baseline SBP 130-139 mmHg and DBP of 89 mmHg or lower or SBP of 139 mmHg or lower and DBP of 85- 89 mmHg, at screening, eligibility and randomization visits
3. Subjects that did not receive any antihypertensive treatment in the past o present
4. Subjects that are willing to sign an informed consent form prior to joining the study

Exclusion Criteria:

1. Subjects with Mean baseline SBP higher than 120 and lower than 130 mmHg
2. Subjects with Mean baseline DBP higher than 80 and lower than 85 mmHg
3. Subjects who are treated for blood pressure reduction (any treatment)
4. Subjects under treatment with other chronic medications (e.g. statins, NSAID etc.)
5. Subjects that use antioxidant agents or vitamins within 4 weeks prior to inclusion into the study
6. Subjects that will not be able to follow the study dietary proscriptions from the screening visit through the final visit
7. Subjects following any special diet including, but not limited to liquid, high or low protein, raw food, vegetarian or vegan, etc
8. Subjects with known allergy to tomatoes, carotenoids, or vitamin E
9. Subjects diagnosed with Diabetes Mellitus
10. Subjects suffering from obesity
11. Subjects Suffering from a clinically significant dyslipidaemia
12. Subjects suffering from cardiac disease; e.g. suffering from cardiac angina, subjects that were diagnosed with and MI, subjects that needed PTCA or CABG. Subjects diagnosed with LVH, CHF or valvular heart disease
13. Subjects diagnosed with PVD
14. Subjects who were diagnosed with Cerebrovascular disease, s/p CVA, TIA
15. Subjects who suffer from any kind of kidney disease
16. Subjects who suffer from chronic liver disease; defined as elevated AST and ALT at least by 2 times of the normal range
17. Subject with history or current use of illegal or "recreational" drugs
18. Subjects with a history of GI disease or surgery within 6 months prior to study inclusion
19. Subjects with a history of malignancy in the past 5 years
20. Subjects with a history of autoimmune disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The effect Lyc-O-Mato on the blood pressure of pre-hypertensive otherwise healthy subjects compared to the placebo group following 12 weeks of treatment | 12 weeks
  Change in blood pressure from baseline to 12 weeks in mmHG

SECONDARY OUTCOMES:
The effect Cardio Mato on the blood pressure of Pre-hypertensive otherwise healthy subjects compared to the placebo group following 4 and 8 weeks of treatment | 4-8 weeks
  Change in blood pressure from baseline to 4 and 8 weeks in mmHG
The correlation between B.P changes in the Cardio Mato or placebo treatment arms during the study with serum lycopene phytofluene, and phytoene levels | 12 weeks
  B.P change

OTHER OUTCOMES:
Number of adverse events recorded during the supplementation period, lycopene compared to placebo | 12 weeks
  AE epizoda

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Aharon, MD., Study Director — LycoRed Ltd.
Locations (1):
- Maccabi Health care, outpatient clinic, Holon, Israel

REFERENCES:
- See also: Data on tomato extracted lycopene — http://www.lycored.com